CLINICAL TRIAL: NCT05624788
Title: A Study to Characterize Access to Specialty Care Received by American Indians/Alaska Natives (CATORI)
Brief Title: A Study to Characterize Access to Specialty Care Received by American Indians/Alaska Natives
Acronym: CATORI
Status: Completed | Type: Observational
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: ML44072
Record Dates: First submitted 2022-11-10; First posted 2022-11-22 (Actual); Last update posted 2025-04-25 (Actual); Status verified 2025-04

CONDITIONS: Specialist Referral: Neurology; Specialist Referral: Ophthalmology; Specialist Referral: Oncology

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Specialist Referral: Neurology
  Interventions: Other: No Intervention
- Specialist Referral: Ophthalmology
  Interventions: Other: No Intervention
- Specialist Referral: Oncology
  Interventions: Other: No Intervention

INTERVENTIONS:
Other: No Intervention — Participants who self-identify as American Indian or Alaska Native with any indication requiring referral to a specialist after a primary care provider standard of care visit will be observed to collect data, using several surveys at 6 and 12 months. No additional specialty care visits will be added for the purpose of this study given the intent to observe medical care received following primary care provider referral. Referral to a specialist will be based on local clinical practice.

SUMMARY:
This is an observational study to define current care pathways for American Indian or Alaska Native patients who require specialty care and potential feasibility of conducting clinical research within the existing framework. The study is designed with the flexibility to enroll patients with any indication requiring referral to one of the following specialists: neurologist, ophthalmologist, or oncologist. Eligible patients will have recently (≤6 months) been referred to a specialty care provider and not yet seen a specialist (in addition to meeting the other eligibility criteria). The PPD virtual site can enroll patients from anywhere across the United States.

The study will collect data to determine whether a patient was seen by a specialist, diagnosed with a specialized disease, patient characteristics potentially associated with being seen or not seen by a specialist, and the reasons/barriers why a patient was not seen by a specialist through a number of patient surveys.

ELIGIBILITY:
Inclusion Criteria:

* Ability to read English at 8th grade proficiency or have a household member willing to assist in translation to complete patient surveys
* Self-identification as American Indian or Alaska Native
* Referred to a neurologist, ophthalmologist, or oncologist for the first time within 6 months of screening and has not been seen by the specialist. Exception: Patients referred to an oncologist who have had a first-time visit with an oncologist but have a pending follow-up visit or pending referral visit within 6 months of screening may be included in the study.
* Personal landline or cell phone and/or access to internet
* Willingness to complete all surveys in the study and participate for 12 months

Exclusion Criteria:

* Currently under the care of a specialist (neurologist, ophthalmologist, or oncologist) to whom they are being referred to by the primary care provider (i.e., to be eligible, the specialty care physician should be new to the participant) at time of screening
* Currently or planned to receive care that requires in participant visits for the indication requiring referral from the primary care provider (e.g., radiotherapy, chemotherapy for cancer diagnosis). Exception: Patients referred to an oncologist who have had a first-time visit with an oncologist but have a pending follow-up visit or pending referral visit may be included in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study will focus exclusively on American Indians and Alaska Native patients who are seen by primary care providers and require an advanced care referral to a specialist.
Sampling Method: Non-Probability Sample
Enrollment: 84 (Actual)
Dates: Start 2022-12-02 (Actual); Primary Completion 2025-04-01 (Actual); Study Completion 2025-04-15 (Actual)

PRIMARY OUTCOMES:
Percentage of All Participants Seen by a Specialist for Advanced Care After Primary Care Provider Referral to a Specialist at 6 Months | 6 Months
Percentage of All Participants Seen by a Specialist for Advanced Care After Primary Care Provider Referral to a Specialist at 12 Months | 12 Months

SECONDARY OUTCOMES:
Percentage of Participants Seen by a Specialist and Treated for Their Disease at 6 Months | 6 Months
Percentage of Participants Seen by a Specialist and Treated for Their Disease at 12 Months | 12 Months
Percentage of Responses by Participant-Reported Barriers to Specialty Referral Completion at 6 Months | 6 Months
Percentage of Responses by Participant-Reported Barriers to Specialty Referral Completion at 12 Months | 12 Months
Percentage of Participants Seen by a Specialist After Primary Care Provider Referral Within Each of the Three Specialist Groups at 6 Months | 6 Months
Percentage of Participants Seen by a Specialist After Primary Care Provider Referral Within Each of the Three Specialist Groups at 12 Months | 12 Months

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Genentech, Inc.
Locations (2):
- United States (2):
  - PPD Virtual - PPD - US, Wilmington, North Carolina
  - Avera Research Institute, Sioux Falls, South Dakota

IPD SHARING:
Plan to Share IPD: No